CLINICAL TRIAL: NCT03872544
Title: Fat to the Future, Dermal Time 3: Short and Medium Term Clinical and Histological Status of Free Dermal Fat Autograft Recipient Sites: Observational Study of a Prospective Cohort Treated for Complex Craniofacial Wounds
Brief Title: Short Term Status of Free Dermal Fat Autografts for Complex Craniofacial Wounds
Acronym: FTFDT3
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dufresne, Craig, MD, PC (Other)
Responsible Party: Sponsor
Other Study IDs: U1111-1229-8480; 000088 (Other: FSRG #1 IRB)
Record Dates: First submitted 2019-03-09; First posted 2019-03-13 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Wound; Head, Multiple; Wound; Head, Scalp; Wound; Head; Wound Infection; Wound Complication; Wound Dehiscence; Wound of Skin; Wound Open; Wounds, Penetrating; Wounds, Nonpenetrating; Wounds and Injuries; Wounds; Disturbance of Wound Healing; Facial Bones Fracture; Soft Tissue Injuries; Skull Fractures; Surgical Wound; Surgical Wound Infection; Wound Healing
Keywords: Autologous Transplantation; Free Tissue Flaps; Graft Survival; Reconstructive Surgical Procedures; Patient Selection; Debridement; Subcutaneous Fat; Surgical Flaps; Treatment Outcome
MeSH Terms: conditions — Wounds and Injuries; Wound Infection; Wounds, Penetrating; Wounds, Nonpenetrating; Soft Tissue Injuries; Skull Fractures; Surgical Wound; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Prepared and stained slides made from the material obtained during biopsies will be retained for use in the clinical care of the patient and research. Other material stored in formalin from biopsy specimens obtained will be banked for future use in immunohistochemistry studies to further define free DFA physiology. Additional IRB approval to use any the material from biopsy specimens for any future studies will be obtained. The specimens will not be shared with outside researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate the use of free autologous dermal fat grafting (also called free dermal fat autografting) to treat complex craniofacial wounds that have failed standard treatment and to understand how well these grafts work to repair wounds long term. Patients who have undergone free autologous dermal fat grafting to treat complex craniofacial wounds less than 1 week ago will have photographs and small biopsies taken of the area that was grafted. Patients will be followed for 2 years to monitor the area that was grafted.

DETAILED DESCRIPTION:
A complex craniofacial wound is a wound on the head or face that will not heal, despite efforts to heal the wound with standard treatments, such as antibiotics and surgery to clean the wound. Currently, there are no good treatment options for these types of complex craniofacial wounds. This study will evaluate what happens when free dermal fat autografting is used to help treat complex craniofacial wounds by evaluating the area where the graft was placed to better understand how these types of grafts function. Free dermal fat autografting is the process of taking fat from under the outer layer of skin and moving it to another part of the body of the same individual. Although free dermal fat autografts have been used for many decades in plastic and reconstructive surgery to help a variety of patients suffering from different problems, only one study has used them to help heal complex craniofacial wounds. This use of free dermal fat autografting is not considered to be experimental or an investigational product by the US Food and Drug Administration (FDA). Still, the use of free dermal fat autografting has not been formally evaluated to understand how these types of grafts help patients with complex craniofacial wounds.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a complex craniofacial wound, defined by failure of initial reconstructive and antibiotic treatment and the presence of chronic infection, exposed hardware, irradiated local tissue, or soft tissue volume loss
* Presence of wound contracture, breakdown of overlying tissue, or challenging anatomical deformities
* Patient has had two or more failed reconstructive attempts or has failed two or more attempts to treat local infection
* Speak, read, and understand English
* Willing to freely give consent
* Is able or has a legal representative to give consent

Exclusion Criteria:

* Absence of a complex craniofacial wound, defined by failure of initial reconstructive and antibiotic treatment and the presence of chronic infection, exposed hardware, irradiated local tissue, or soft tissue volume loss
* Absence of wound contracture, breakdown of overlying tissue, or challenging aesthetic deformities
* Patient has not had two or more failed reconstructive attempts or has not failed two or more attempts to treat local infection
* Does not speak, read, or understand English
* Unwilling to freely give consent
* Is unable or does not have a legal representative to give consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential patients are any consecutive patients not part of a retrospective cohort who undergo free autologous dermal fat grafting for one or more complex craniofacial wounds, carried out by a single sub-speciality trained plastic surgeon (Study Principal Investigator).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
Change in drainage, erythema, oedema, and pain; and the presence of intact tissues associated with the wound | Evaluated through study completion, an average of 2 years.
  Visually appraised evidence of drainage, erythema, oedema, and pain; and the presence of intact tissues associated with the wound

SECONDARY OUTCOMES:
Change in volume and contour of the defect associated with the wound | Evaluated through study completion, an average of 2 years.
  Visually appraised volume and contour of the defect associated with the wound
Concentration of adipocytes, mast cells, macrophages, and dermal lymphocytes in the wound site | Evaluated through study completion, an average of 2 years.
Ratio for tissue type in the wound site | Evaluated through study completion, an average of 2 years.
  Tissue types considered are adipose and fibrous.
Ratio of immune cell populations in the wound site | Evaluated through study completion, an average of 2 years.
  Immune cell types considered are mast cells, macrophages, and dermal lymphocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Dufresne, MD, Principal Investigator — Dr Craig R Dufresne, MD, PC
Locations (1):
- Office of Craig R Dufresne, MD, PC, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) or biospecimens will be shared.

REFERENCES:
- [Background] Dufresne CR, Poling MI. Free Dermal Fat Autografting for Complex Craniofacial Wounds. J Craniofac Surg. 2020 Sep;31(6):1563-1567. doi: 10.1097/SCS.0000000000006398. PMID 32310868
- [Background] Dufresne CR, Poling MI. Free Dermal Fat Autografts for Complex Craniofacial Wounds: A 3-decade, Retrospective Cohort Study. PRS Global Open. 2019 August; 7(8S-1):101. doi: 10.1097/01.GOX.0000584800.01063.18.
- See also: Principal Investigator's (Dr Craig R Dufresne) Research and Press Relations main webpage. Last Accessed: 7 Jun 2022 — https://www.duplastics.com/research-press/